CLINICAL TRIAL: NCT03767192
Title: A Multicenter, Randomized, Double Blind, Sham Control, Parallel Arm Trial to Assess Effectiveness and Safety of the Ischemic Stroke System ISS, as an Adjunct to Standard of Care in Subjects With Acute Ischemic Stroke
Brief Title: Implant for Augmentation of Cerebral Blood Flow Trial, Effectiveness and Safety in a 24 Hour Window (ImpACT-24A)
Acronym: ImpACT-24A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol Amendment
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLP1000500-24A
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; randomized clinical trial; effectiveness; safety
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Stimulation (Experimental): Device: The Ischemic Stroke System SPG stimulation and standard of care
  Interventions: Device: Active Stimulation
- Sham Stimulation (Sham Comparator): Device: Sham control Sham stimulation and standard of care
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Active Stimulation — SPG stimulation and standard of care
  Arms: Active Stimulation
Device: Sham Stimulation — Sham SPG stimulation and standard of care
  Arms: Sham Stimulation

SUMMARY:
The primary objective of the study is to assess the safety and effectiveness of SPG stimulation with the ISS in patients with an acute ischemic stroke in the anterior circulation initiated within 24 hours from stroke onset.

DETAILED DESCRIPTION:
This study was first registered as NCT00826059 on January 19, 2009 under the name ImpACT-24.

Background:

Recruitment to ImpACT-24 was halted, the protocol was amended and then the study was resumed. Later, it was decided to define the first part (before the halt) as a separate study - ImpACT-24A, and identify the continuation of the study as ImpACT-24B. ImpACT-24B continues to be registered as NCT00826059, and ImpACT-24A is registered in this new record.

Detailed Description:

A multi-center, multinational, randomized, double blind, sham control, adjunctive to Standard of Care, parallel arm study with ongoing DSMB review of accumulated safety data.

Screening:

Treatment should be initiated between 8 and 24 hours from stroke onset. All screened patients will be identified by patient number and will sign the informed consent prior to any study procedure initiation.

Period 1: Day 1-5

Day 1- Eligible subjects will be randomized in a 2:1 (ISS Stimulation: Sham Control) ratio:

Group 1: Implantation and ISS Stimulation during five consecutive days & Standard of Care Group 2: Implantation and Sham Stimulation during five consecutive days & Standard of Care The implantation will be performed by a trained physician. Stimulation/sham stimulation will be delivered Day 2-5 ISS / Sham Stimulation will be repeated during the following four consecutive days by trained personnel within 18-26 hours from preceding stimulation.

Day 5 / Day of Discharge. Following the last ISS /Sham Stimulation, explantation will be performed.

Subjects will continue with Standard of Care as needed and will be released from the hospital upon investigator's judgment.

Period 2: Day of Discharge - 90±7 days During this period both groups (ISS Stimulation and Sham Control) will be treated according to Standard of Care either at the hospital, rehabilitation center or at home.

Scheduled visits will be performed on day 30±7 and day 60 ±7, which will include safety and effectiveness assessments.

Final Visit Day 90±7 days: The final visit will be performed at the study site and will include safety and effectiveness evaluations.

Patients will be contacted by study personnel via telephone on Day 180±7 and on Day 360±7 in order to assess their quality of life status.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years and ≤ 85 of both genders.
2. Clinical diagnosis of an acute ischemic stroke in the Carotid, Middle or Anterior Cerebral Artery territories
3. Baseline NIHSS ≥ 7 and ≤ 18
4. Ability to initiate treatment within 8- 24 hours from stroke onset.

Exclusion Criteria:

1. Intracranial hemorrhage or hemorrhagic transformation
2. Massive stroke
3. Acute ischemic stroke in the posterior circulation
4. Minor stroke
5. Treated with IV-tPA ,IA-tPA or neurothrombectomy devices for the current stroke
6. Previous stroke in the last 6 months or pre-existing disability
7. Patients with bleeding propensity or any condition in the oral cavity that prevents implantation
8. Known cerebral arteriovenous malformation, cerebral aneurysm.
9. Clinical suspicion of septic embolus.
10. Uncontrolled hypertension (systolic >185 mmHg and/or diastolic >110 mmHg)
11. Serious systemic infection.
12. Women known to be pregnant or having a positive or indeterminate pregnancy test.
13. Patients with other implanted neural stimulator/ electronic devices (pacemakers).
14. Life expectancy < 1 year from causes other than stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Sliding Dichotomy modified Rankin Scale (mRS) at 3 months | 90 ±7 days
  Final global disability level on the modified Rankin scale (mRS) at 3 months better than expectation (sliding dichotomy analysis) ) assessed in the modified intention to treat (mITT) population defined as all randomized subjects receiving at least the minimal exposure of 1 treatment (ISS Stimulation or Sham Control) session out of the 5 planned sessions.
  mRS Scale:
  * 0 - No symptoms.
  * 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
  * 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * 3 - Moderate disability. Requires some help, but able to walk unassisted.
  * 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * 6 - Dead.
Number of participants with Serious Adverse Events | 90 ±7 days
  Comparison between the active and sham stimulation groups of all serious adverse events (SAEs)
Number of participants with neurological deterioration | 10 days
  Comparison between the active and sham stimulation groups of the rate of neurological deterioration, defined as an increase of 4 or more points on the NIHSS related to any neurological event within the first 10 days after stroke onset
Number of participants with implantation complications | 90 ±7 days
  The rate of implantation complications as classified by the investigator
Number of participants with stimulation-related adverse events | 90 ±7 days
  Comparison between the active and sham stimulation groups of stimulation-related adverse events as classified by the investigator
Mortality rate | 90 ±7 days
  Comparison of mortality rates between the active and sham stimulation groups

SECONDARY OUTCOMES:
Sliding Dichotomous 90-day mRS for patients with Aphasia at baseline | 90 ±7 days
  Sliding Dichotomous 90-day mRS for patients with Aphasia at baseline
  mRS Scale:
  * 0 - No symptoms.
  * 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
  * 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * 3 - Moderate disability. Requires some help, but able to walk unassisted.
  * 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * 6 - Dead.
Binary NIHSS at Day 90 | 90 ±7 days
  Binary NIHSS (success for score ≤1 or for ≥ 9-point improvement versus baseline)
  The NIHSS (National Institute of Health Stroke Score) is a 42-point scale that quantifies neurological deficits in 11 categories. Ratings for each item are scored with 3 to 5 grades, with 0 as normal.
Stroke-related quality of life at 3 months: Stroke Impact Scale-16 | 90 ±7 days
  Stroke-related quality of life at 3 months according to the Stroke Impact Scale-16 (SIS-16)
  The scale is based on a questionnaire with 16 items. Each answer ranges from 1 (poor) to 5 (good). A final single-item Recovery domain assesses the individual's perception of his/her recovery from stroke, where:
  0 = no recovery 100 = full recovery.
  Domain scores range from 0-100 and are calculated using the following equation:
  Domain score = [(Mean item score - 1) / (5-1) ] x 100

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shay, Study Director — BrainsGate
Locations (8):
- Erlanger Stroke Center, Chattanooga, Tennessee, United States
- Germany (5):
  - Erlangen University Clinic, Erlangen
  - Essen University Clinic, Essen
  - Heidelberg University Clinic, Heidelberg
  - Leipzig University Clinic, Leipzig
  - Munster University Clinic, Münster
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona, Girona

REFERENCES:
- [Derived] Bornstein NM, Saver JL, Diener HC, Gorelick PB, Shuaib A, Solberg Y, Devlin T, Leung T, Molina CA; ImpACT-24A Investigators. Sphenopalatine Ganglion Stimulation to Augment Cerebral Blood Flow: A Randomized, Sham-Controlled Trial. Stroke. 2019 Aug;50(8):2108-2117. doi: 10.1161/STROKEAHA.118.024582. Epub 2019 May 23. PMID 31117920